CLINICAL TRIAL: NCT05181319
Title: Development of a Nomogram for Predicting Bronchopulmonary Dysplasia in Infants
Brief Title: Prediction for Bronchopulmonary Dysplasia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Kai Mu (Other)
Responsible Party: Sponsor-Investigator, Kai Mu, professor, Qianfoshan Hospital
Organization: Qianfoshan Hospital (Other)
Other Study IDs: QFS-2018-1201
Record Dates: First submitted 2021-12-18; First posted 2022-01-06 (Actual); Last update posted 2022-01-06 (Actual); Status verified 2021-12

CONDITIONS: Bronchopulmonary Dysplasia
Keywords: Bronchopulmonary Dysplasia; Infants；Nomogram
MeSH Terms: conditions — Bronchopulmonary Dysplasia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- bronchopulmonary dysplasia group: infants diagnosed with bronchopulmonary dysplasia
  Interventions: Other: occurrence of bronchopulmonary dysplasia
- no bronchopulmonary dysplasia: infants not diagnosed with bronchopulmonary dysplasia
  Interventions: Other: occurrence of bronchopulmonary dysplasia

INTERVENTIONS:
Other: occurrence of bronchopulmonary dysplasia — We observe the incidence of bronchopulmonary dysplasia

SUMMARY:
In this Multi-center study performed from January 2018, we reviewed data on infants whose gestational ages were below 36 weeks. we collected data containing maternal diseases and neonatal clinical features. LASSO regression was used to select variables for the risk model. Then, we used multivariable logistic regression to build the prediction model incorporating these selected features. Discrimination was assessed by the C-index, and and calibration of the model was assessed by and calibration curve and the Hosmer-Lemeshow test.

ELIGIBILITY:
Inclusion Criteria:

* Patients were recruited from Multi-center Collaborative Group Hospital Neonatal Intensive Care Unit (NICU) Department.
* Patients with gestational age <36 weeks
* admitted to the NICU within 24 h after birth
* the length of stay was more than 1 week

Exclusion Criteria:

* patients with inherited disease, metabolic disorders and multiple malformations.

Max Age: 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Patients were recruited from Multi-center Collaborative Group Hospital Neonatal Intensive Care Unit (NICU) Department. The data was collected from medical records. Patients with GAs <36 weeks, and who were admitted to the NICU within 24 h after birth were included, and the length of stay was more than 1 week.patients with inherited disease, metabolic disorders and multiple malformations were excluded.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
bronchopulmonary dysplasia occurs | 2 weeks after admission
  Number of cases of bronchopulmonary dysplasia

CONTACTS AND LOCATIONS:
Overall Officials: MU Kai, Doctor, Study Director — Qianfoshan Hospital
Locations (1):
- Qianfoshan Hospital, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: No